CLINICAL TRIAL: NCT05670132
Title: Impact of a Neuro-cardiac Rehabilitation Program on the Quality of Life of Children, Adolescents, and Young Adults With Congenital Heart Disease: the Multicentre Randomized Controlled QUALINEUROREHAB Trial
Brief Title: Neuro-cardiac Rehabilitation in Youth With Congenital Heart Disease (QUALINEUROREHAB)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2021/66
Record Dates: First submitted 2022-12-19; First posted 2023-01-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Congenital Heart Disease
Keywords: Neuro-cardiac rehabilitation program; Quality of life
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurocardiac rehabilitation program (Experimental): The home-based neuro-cardiac rehabilitation program will consist of weekly sessions of neuro-cardiac training during 12 weeks at home.
  * The physical activity training consists of two 1-hour sessions of adapted physical activities per week supervised by an APA educator or equal. One weekly session is held in person, at home, and the second one in videoconference. All training sessions follow the same scheme with 30 minutes of bicycle training, adapted from high-intensity training (30-33), and 30 minutes of "free" adapted physical activities
  * The neuropsychological component will consist of 2 home-based weekly 25-minute sessions of computerized cognitive training via the new platform of CogMed (standard format) for the patient and 1 weekly 30/45-min teleconsultation session of neuropsychological feedback on every-day life emotional regulation and executive functioning applied to school and family life for either the parent (for ages 17 and younger) or young adults with CHD.
  Interventions: Other: Neurocardiac rehabilitation program
- Standard of care (Active Comparator): The control group will follow European recommendations for cardiology care (standard of care) without introducing any additional interventions for research purposes at the exception of primary (HRQoL questionnaires) and secondary outcomes
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Neurocardiac rehabilitation program — Patients receiving a neurocardiac rehabilitation program for 12 weeks.
  Arms: Neurocardiac rehabilitation program
Other: Standard of care — No intervention during the neurocardiac rehabilitation program
  Arms: Standard of care

SUMMARY:
Remarkable progress in paediatric cardiology and surgery have led to the substantial increase of congenital heart disease (CHD) survivors. Long-term outcomes in rare and complex CHD have become a critical priority as three major sources of morbidity have been identified in this population: neurodevelopmental sequelae, mental health issues and reduced exercise capacity. These challenges adversely affect their quality of life and constitute a major public health issue. We seek to evaluate the efficacy of the first integrative and holistic program in Neuro-Cardiac Health associating physical and psychological rehabilitation for children with rare CHD compared to the standard of care. Children randomly assigned to the intervention will undergo a 12-week neuro-cardiac intervention including home-based adaptive physical exercise, telehealth parent and child psycho-education and child computerized cognitive training, as well in-person individual sessions of intervention reinforcement. Parents will be actively involved and will receive personalized feedback and educational resources. Children assigned to the control group will receive the standard of care in congenital cardiology. Post-intervention effects will be measured after 12-months on several outcomes including health-related quality of life (HRQoL), trained and untrained cognitive skills, mental health outcomes and cardiovascular/physical variables.

DETAILED DESCRIPTION:
Neurodevelopmental and mental health issues and reduced exercise capacity are the most frequent long-term morbidities in youth with CHD. These problems worsen with age and play a critical role in reducing the quality of life of patients and their families. The QUALI-NEUROREHAB CHD multicentre, randomized controlled trial seeks to test the efficacy of an innovative home-based neuro-cardiac intervention to improve physical and mental health of children, adolescents and young adults with rare CHD, as assessed by the patients themselves using patient-reported outcomes and standardized assessments. Outcomes relate to changes in scores for health-related quality of life (HRQoL, primary outcome measure), neurodevelopmental and mental health outcomes, and cardiopulmonary exercise test parameters, 12 months post-enrolment, in patients with rare CHD aged 8 to 25 years old. This is a two-arm parallel design study: intervention versus control. Intervention using the neuro-cardiac rehabilitation program will be the active arm. Standard of care will be used for the control group and involves normal cardiology consultations and follow-up without intervention programs on physical activity or neurocognitive training. The intervention group will include 12 weeks of neuro-cardiac training, comprised of at-home adaptive physical exercise, telehealth consultations and computerized neurocognitive training as well in-person individual sessions of intervention reinforcement. We hypothesize an increase in the overall HRQoL score of 6 ± 14 points (over 100). With a 90% power, a bilateral alpha risk of 5%, and potentially 20% of loss to follow-up and/or missing data on the primary outcome, we need to randomize 145 patients to each group (N= 290, overall). Analysis will be performed using intent to treat (ITT) approach. We predict significant positive changes in quality of life, mental and physical health scores in patients who will be assigned to the neuro-cardiac intervention (active arm). If this intervention is effective, it can have critical public health implications for the organization and modalities of care for children with rare CHD in Europe. A neuro-cardiac rehabilitation programme tailored to the specific challenges of individuals with rare CHD would improve patient care pathways across major centers in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a CHD of moderate to great complexity as defined in the 2019 AHA/ACC guidelines (Appendix 2)85.
2. History of cardiac surgery and/or catheter-based cardiac intervention(s) during the first year of life.
3. Age between 8 and 25 years at the time of enrolment.
4. Parental or legal guardian's consent for minors (<18 years) and personal consent for adults.
5. Social security affiliation (for France only)

Exclusion Criteria:

1. Unstable and/or severe heart failure: severe heart failure (class IV NYHA functional class), recent decompensated heart failure requiring hospitalisation and/or any significant change in medication (< 3 months before enrolment), systolic ventricle dysfunction (left ventricle or systemic ventricle ejection fraction < 50%)82.
2. Severe hypoxaemia: pulse oxygen saturation (SpO2) at rest <85%, and/or SpO2 at exercise <80%, and/or patient requiring oxygen therapy.
3. Pulmonary hypertension as defined by the 2020 ESC guidelines, whatever the aetiology83.
4. Significant systolic right ventricle (sRV) hypertension (sRV pressure > 50% of systemic systolic pressure).
5. Uncontrolled arrhythmia: symptomatic treated or untreated arrhythmia at rest and/or exercise, treated arrhythmia with sustained supraventricular or ventricular tachycardia on ECG monitoring or during exercise and/or CPET, occurrence or aggravation of any supraventricular or ventricular arrhythmia during exercise and/or CPET.
6. Advanced atrioventricular block (degree 2 or 3), occurrence or aggravation of any conduction disorder during exercise and/or CPET.
7. Uncontrolled arterial hypertension at rest (e.g. if the blood pressure at rest during the consultation >140/90 mmHg in adults, >95th percentile in children84).
8. Acute or recent (< 3 months) myocarditis and pericarditis.
9. Symptomatic aortic or sub-aortic stenosis (mean gradient > 50 mmHg).
10. Non-corrected coarctation of the aorta (surgical or catheter-based repair) with a clinical systolic gradient > 20 mmHg.
11. Dilatation of the aorta (aortic root > 40 mm in adults, > 2 Z-score in children85 (http://www.parameterz.com/sites/aortic-root) except in the case of repaired congenital heart disease with dilatation of the aorta inherent in the malformation and without risk of aortic dissection (tetralogy of Fallot, pulmonary atresia with IVC, common trunk artery).
12. Severe hypertrophic obstructive cardiomyopathy.
13. Acute systemic illness.
14. Recent (<3 months) intracardiac thrombus, embolism, or thrombophlebitis.
15. Inability to follow instructions and/or complete the questionnaires, as determined by the investigator.
16. Absolute contraindications for CPET: fever, uncontrolled asthma, respiratory failure, acute myocarditis or pericarditis, uncontrolled arrhythmias causing symptoms or haemodynamic compromise, uncontrolled heart failure, acute pulmonary embolus or pulmonary infarction, and patients with mental impairment leading to inability to cooperate.
17. Inability to undergo the physical intervention: inability to physically exercise, any invasive medical intervention occurring within 6 months preceding the enrolment or scheduled during the 12-month study period (such as cardiac surgery, catheter-based intervention, orthopaedic surgery, chemotherapy for cancer, or any other significant medical treatment or intervention, as determined by the investigator).
18. Patient with a previously diagnosed severe psychiatric disorder requiring hospitalization and/or continuous specialized care by a psychiatrist, as determined by the investigator.
19. Patients who benefited from a cardiac rehabilitation within the 12 months preceding the enrolment.
20. Patients who benefited from a computerized executive function or attention training such as Cogmed Working Memory Program within the 12 months preceding the enrolment.
21. For female patients: pregnancy, pregnancy plan, or breastfeeding woman following questioning of the patient.
22. Patients deprived of liberty due to an ongoing legal procedure, adult's patient under guardianship or curatorship or unable to personally express their consent.
23. Any other clinical and/or pharmacological treatment that is believed to interfere with the study or the optimal clinical care.
24. Initiation or total withdrawal of psychotropic medication (i.e., any psychotropic medication including methylphenidate, benzodiazepines, and mood stabilizers) within the 6 months preceding the enrolment.
25. Patient participating or wishing to participate in any interventional clinical research (drug trial, medical device, non-drug trial).

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2027-06-03 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Total score of the Pediatric Quality of Life Inventory (PedsQL) 4.0 questionnaire | between Month 0 and Month 12
  Change in the self-reported total score of the PedsQL 4.0 questionnaire between baseline (Month 0) and the end of follow-up (Month 12) in both groups.

SECONDARY OUTCOMES:
Proxy-reported total score of the Pediatric Quality of Life Inventory (PedsQL) for paediatric patients | between Month 0 and Month 12
Pediatric Quality of Life Inventory (PedsQL) 4.0 Health-related quality (HRQoL ) of life questionnaire score per dimension (self and proxy reports) | between Month 0 and Month 12
Behaviour Rating Inventory of Executive Function (BRIEF) scale scores | between Month 0 and Month 12
  BRIEF (8-18 years) and BRIEF-A (older than 18 years)
  These scales make it possible to identify executive dysfunctions that have an impact on daily life.
  BRIEF assesses behaviours based on questions grouped into 8 scales: inhibition, flexibility, emotional control, initiation, material organization, working memory, planning/organization, and control.
  For the BRIEF-A (18 years and +), 9 scales are available and those yield the same indices and general composite score.
Wisconsin Card Sorting Test scale score | between Month 0 and Month 12
  This test measures higher-order executive functioning including planning, anticipation, and cognitive flexibility.
Wechsler Intelligence Scale scores | between Month 0 and Month 12
  Scores on the main indices of the Wechsler Intelligence Scale (WISC-V for children, WAIS-IV for adults): verbal comprehension, visual-spatial abilities, working memory, fluid reasoning and processing speed.
NEPSY-II scale scores | between Month 0 and Month 12
  Score on tests of language (comprehension of instructions) and social cognition (understanding of facial emotions and theories of mind) from the NEPSY-II Child Neuropsychological Assessment battery
Wechsler Adult Memory Scale scores | between Month 0 and Month 12
  verbal and visual memory tests
Vineland questionnaire | between Month 0 and Month 12
  The Vineland-2 proxy-questionnaire of adaptive functioning: this is a parent- or other informant report on adaptive skills including social, communication, academic and daily-life independence of children.
Multiscore Depression Inventory for Children (MDI-C) scale score | between Month 0 and Month 12
  Scale providing access to the child's emotional world and more specifically to depression through 8 dimensions: self-esteem, anxiety, sad mood, social introversion, pessimism, defiance, low energy, and feelings of powerlessness.
Beck's Depression Inventory (BDI) scale score | between Month 0 and Month 12
  Self-report questionnaire (BDI-2) used to measure the characteristic attitudes and symptoms of depression
Revised Child Manifest Anxiety Scale (R-CMAS) score | between Month 0 and Month 12
  Self-administered questionnaire providing a more specific assessment of anxiety in its multiple expressions: worry/hypersensitivity, physiological anxiety, and social concern/concentration, based on a global measure of the child's or adolescent's anxiety level.
State-Trait Anxiety Inventory (STAI) - Form Y score | between Month 0 and Month 12
Resilience Scale score | between Month 0 and Month 12
  Resilience Scale for Children (RS10) score and Resilience Scale for Adults: self-administered questionnaire relating to the ability to cope and respond to life events.
Cardiopulmonary exercise test (CPET) | between Month 0 and Month 12
Muscular strength | between Month 0 and Month 12
  Muscular strength measured using a handgrip dynamometer . This parameter represents the strength of the upper extremities and correlates with inspiratory muscle function and Vital Capacity (FVC) of the lungs. It is measured three times on both hands while sitting with the elbows in a rectangular position. The highest value of the better arm will be used.
Metabolic equivalent of task (MET) | between Month 0 and Month 12
  Physical activity intensity and energy expenditure measured by an actimeter
Following physical activity questionnaires | between Month 0 and Month 12
  Self-administrated questionnaire : International Physical Activity Questionnaire(IPAQ) for patients ≥18 years
Following physical activity questionnaires | between Month 0 and Month 12
  Self-administrated questionnaire : Physical Activity Questionnaire for Children (PAQ-C) for 14 to 17-year-old children
Following physical activity questionnaires | between Month 0 and Month 12
  Self-administrated questionnaire : Physical Activity Questionnaire for Children (PAQ-A) for 8 to 14-year-old children

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD,PhD, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- Saint-Luc University Hospital, Brussels, Belgium
- France (3):
  - University Hospital of Montpellier - Arnaud de Villeneuve Hospital, Montpellier
  - Saint-Pierre Institute, Palavas-les-Flots
  - University Hospital of Bordeaux - Haut-Levêque Hospital, Pessac
- Deutsches Herzzentrum München, München, Germany

REFERENCES:
- [Background] Amedro P, Dorka R, Moniotte S, Guillaumont S, Fraisse A, Kreitmann B, Borm B, Bertet H, Barrea C, Ovaert C, Sluysmans T, De La Villeon G, Vincenti M, Voisin M, Auquier P, Picot MC. Quality of Life of Children with Congenital Heart Diseases: A Multicenter Controlled Cross-Sectional Study. Pediatr Cardiol. 2015 Dec;36(8):1588-601. doi: 10.1007/s00246-015-1201-x. Epub 2015 May 31. PMID 26024647
- [Background] Muller J, Christov F, Schreiber C, Hess J, Hager A. Exercise capacity, quality of life, and daily activity in the long-term follow-up of patients with univentricular heart and total cavopulmonary connection. Eur Heart J. 2009 Dec;30(23):2915-20. doi: 10.1093/eurheartj/ehp305. Epub 2009 Aug 18. PMID 19692392
- [Background] Amedro P, Picot MC, Moniotte S, Dorka R, Bertet H, Guillaumont S, Barrea C, Vincenti M, De La Villeon G, Bredy C, Soulatges C, Voisin M, Matecki S, Auquier P. Correlation between cardio-pulmonary exercise test variables and health-related quality of life among children with congenital heart diseases. Int J Cardiol. 2016 Jan 15;203:1052-60. doi: 10.1016/j.ijcard.2015.11.028. Epub 2015 Nov 10. PMID 26638054
- [Background] Amedro P, Gavotto A, Guillaumont S, Bertet H, Vincenti M, De La Villeon G, Bredy C, Acar P, Ovaert C, Picot MC, Matecki S. Cardiopulmonary fitness in children with congenital heart diseases versus healthy children. Heart. 2018 Jun;104(12):1026-1036. doi: 10.1136/heartjnl-2017-312339. Epub 2017 Nov 23. PMID 29170358
- [Background] Muller J, Bohm B, Semsch S, Oberhoffer R, Hess J, Hager A. Currently, children with congenital heart disease are not limited in their submaximal exercise performance. Eur J Cardiothorac Surg. 2013 Jun;43(6):1096-100. doi: 10.1093/ejcts/ezs712. Epub 2013 Jan 22. PMID 23345176
- [Background] Calderon J, Bellinger DC, Hartigan C, Lord A, Stopp C, Wypij D, Newburger JW. Improving neurodevelopmental outcomes in children with congenital heart disease: protocol for a randomised controlled trial of working memory training. BMJ Open. 2019 Feb 19;9(2):e023304. doi: 10.1136/bmjopen-2018-023304. PMID 30782877
- [Background] Calderon J, Angeard N, Moutier S, Plumet MH, Jambaque I, Bonnet D. Impact of prenatal diagnosis on neurocognitive outcomes in children with transposition of the great arteries. J Pediatr. 2012 Jul;161(1):94-8.e1. doi: 10.1016/j.jpeds.2011.12.036. Epub 2012 Jan 28. PMID 22284567
- [Background] Calderon J, Stopp C, Wypij D, DeMaso DR, Rivkin M, Newburger JW, Bellinger DC. Early-Term Birth in Single-Ventricle Congenital Heart Disease After the Fontan Procedure: Neurodevelopmental and Psychiatric Outcomes. J Pediatr. 2016 Dec;179:96-103. doi: 10.1016/j.jpeds.2016.08.084. Epub 2016 Sep 28. PMID 27692462
- [Background] Pelliccia A, Sharma S, Gati S, Back M, Borjesson M, Caselli S, Collet JP, Corrado D, Drezner JA, Halle M, Hansen D, Heidbuchel H, Myers J, Niebauer J, Papadakis M, Piepoli MF, Prescott E, Roos-Hesselink JW, Graham Stuart A, Taylor RS, Thompson PD, Tiberi M, Vanhees L, Wilhelm M; ESC Scientific Document Group. 2020 ESC Guidelines on sports cardiology and exercise in patients with cardiovascular disease. Eur Heart J. 2021 Jan 1;42(1):17-96. doi: 10.1093/eurheartj/ehaa605. No abstract available. PMID 32860412
- [Background] Amedro P, Gavotto A, Legendre A, Lavastre K, Bredy C, De La Villeon G, Matecki S, Vandenberghe D, Ladeveze M, Bajolle F, Bosser G, Bouvaist H, Brosset P, Cohen L, Cohen S, Corone S, Dauphin C, Dulac Y, Hascoet S, Iriart X, Ladouceur M, Mace L, Neagu OA, Ovaert C, Picot MC, Poirette L, Sidney F, Soullier C, Thambo JB, Combes N, Bonnet D, Guillaumont S. Impact of a centre and home-based cardiac rehabilitation program on the quality of life of teenagers and young adults with congenital heart disease: The QUALI-REHAB study rationale, design and methods. Int J Cardiol. 2019 May 15;283:112-118. doi: 10.1016/j.ijcard.2018.12.050. Epub 2018 Dec 20. PMID 30616811
- [Background] Calderon J, Wypij D, Rofeberg V, Stopp C, Roseman A, Albers D, Newburger JW, Bellinger DC. Randomized Controlled Trial of Working Memory Intervention in Congenital Heart Disease. J Pediatr. 2020 Dec;227:191-198.e3. doi: 10.1016/j.jpeds.2020.08.038. Epub 2020 Aug 19. PMID 32827526
- [Background] Meyer M, Brudy L, Fuertes-Moure A, Hager A, Oberhoffer-Fritz R, Ewert P, Muller J. E-Health Exercise Intervention for Pediatric Patients with Congenital Heart Disease: A Randomized Controlled Trial. J Pediatr. 2021 Jun;233:163-168. doi: 10.1016/j.jpeds.2021.01.058. Epub 2021 Jan 29. PMID 33516681
- [Background] Abassi H, Gavotto A, Picot MC, Bertet H, Matecki S, Guillaumont S, Moniotte S, Auquier P, Moreau J, Amedro P. Impaired pulmonary function and its association with clinical outcomes, exercise capacity and quality of life in children with congenital heart disease. Int J Cardiol. 2019 Jun 15;285:86-92. doi: 10.1016/j.ijcard.2019.02.069. Epub 2019 Mar 1. PMID 30857849
- [Background] Morales Mestre N, Reychler G, Goubau C, Moniotte S. Correlation Between Cardiopulmonary Exercise Test, Spirometry, and Congenital Heart Disease Severity in Pediatric Population. Pediatr Cardiol. 2019 Apr;40(4):871-877. doi: 10.1007/s00246-019-02084-5. Epub 2019 Mar 8. PMID 30850878
- [Background] Hager A, Hess J. Comparison of health related quality of life with cardiopulmonary exercise testing in adolescents and adults with congenital heart disease. Heart. 2005 Apr;91(4):517-20. doi: 10.1136/hrt.2003.032722. PMID 15772218
- [Background] Muller J, Berner A, Ewert P, Hager A. Reduced health-related quality of life in older patients with congenital heart disease: a cross sectional study in 2360 patients. Int J Cardiol. 2014 Aug 1;175(2):358-62. doi: 10.1016/j.ijcard.2014.06.008. Epub 2014 Jun 18. PMID 24973809
- [Background] Amedro P, Bajolle F, Bertet H, Cheurfi R, Lasne D, Nogue E, Auquier P, Picot MC, Bonnet D. Quality of life in children participating in a non-selective INR self-monitoring VKA-education programme. Arch Cardiovasc Dis. 2018 Mar;111(3):180-188. doi: 10.1016/j.acvd.2017.05.013. Epub 2017 Nov 1. PMID 29100908
- [Background] Werner O, Abassi H, Lavastre K, Guillaumont S, Picot MC, Serrand C, Dulac Y, Souletie N, Acar P, Bredy C, Amedro P. Factors influencing the participation of adolescents and young adults with a congenital heart disease in a transition education program: A prospective multicentre controlled study. Patient Educ Couns. 2019 Dec;102(12):2223-2230. doi: 10.1016/j.pec.2019.06.023. Epub 2019 Jun 26. PMID 31262673
- [Background] Abassi H, Bajolle F, Werner O, Auer A, Marquina A, Mura T, Lavastre K, Guillaumont S, Manna F, Auquier P, Bonnet D, Amedro P. Health-related quality of life correlates with time in therapeutic range in children on anticoagulants with International Normalised Ratio self-monitoring. Arch Cardiovasc Dis. 2020 Dec;113(12):811-820. doi: 10.1016/j.acvd.2020.05.022. Epub 2020 Oct 14. PMID 33069639
- [Background] Abassi H, Huguet H, Picot MC, Vincenti M, Guillaumont S, Auer A, Werner O, De La Villeon G, Lavastre K, Gavotto A, Auquier P, Amedro P. Health-related quality of life in children with congenital heart disease aged 5 to 7 years: a multicentre controlled cross-sectional study. Health Qual Life Outcomes. 2020 Nov 12;18(1):366. doi: 10.1186/s12955-020-01615-6. PMID 33183312
- [Background] Amedro P, Gavotto A, Bredy C, Guillaumont S. [Cardiac rehabilitation for children and adults with congenital heart disease]. Presse Med. 2017 May;46(5):530-537. doi: 10.1016/j.lpm.2016.12.001. Epub 2017 Jan 23. French. PMID 28126509
- [Background] Calderon J, Newburger JW. Working Memory Training: A Promising Intervention? Crit Care Med. 2018 Jul;46(7):1199-1201. doi: 10.1097/CCM.0000000000003172. No abstract available. PMID 29912106
- [Background] Moreau J, Lavastre K, Romieu H, Charbonnier F, Guillaumont S, Bredy C, Abassi H, Werner O, De La Villeon G, Requirand A, Auer A, Matecki S, Karsenty C, Guitarte A, Hadeed K, Dulac Y, Souletie N, Acar P, Bajolle F, Bonnet D, Negre-Pages L, Mura T, Mounier M, Seguela PE, Thomas J, Iriart X, Jean-Benoit-Thambo, Amedro P. Impact of Sophrology on cardiopulmonary fitness in teenagers and young adults with a congenital heart disease: The SOPHROCARE study rationale, design and methods. Int J Cardiol Heart Vasc. 2020 Mar 3;27:100489. doi: 10.1016/j.ijcha.2020.100489. eCollection 2020 Apr. PMID 32154361
- [Background] Amedro P, Werner O, Abassi H, Boisson A, Souilla L, Guillaumont S, Calderon J, Requirand A, Vincenti M, Pommier V, Matecki S, De La Villeon G, Lavastre K, Lacampagne A, Picot MC, Beyler C, Delclaux C, Dulac Y, Guitarte A, Charron P, Denjoy-Urbain I, Probst V, Baruteau AE, Chevalier P, Di Filippo S, Thambo JB, Bonnet D, Pasquie JL. Health-related quality of life and physical activity in children with inherited cardiac arrhythmia or inherited cardiomyopathy: the prospective multicentre controlled QUALIMYORYTHM study rationale, design and methods. Health Qual Life Outcomes. 2021 Jul 28;19(1):187. doi: 10.1186/s12955-021-01825-6. PMID 34321045
- [Background] Gavotto A, Huguet H, Picot MC, Guillaumont S, Matecki S, Amedro P. The V̇e/V̇co2 slope: a useful tool to evaluate the physiological status of children with congenital heart disease. J Appl Physiol (1985). 2020 Nov 1;129(5):1102-1110. doi: 10.1152/japplphysiol.00520.2020. Epub 2020 Sep 10. PMID 32909919
- [Background] Werner O, Bredy C, Lavastre K, Guillaumont S, De La Villeon G, Vincenti M, Gerl C, Dulac Y, Souletie N, Acar P, Pages L, Picot MC, Bourrel G, Oude Engberink A, Million E, Abassi H, Amedro P. Impact of a transition education program on health-related quality of life in pediatric patients with congenital heart disease: study design for a randomised controlled trial. Health Qual Life Outcomes. 2021 Jan 19;19(1):23. doi: 10.1186/s12955-021-01668-1. PMID 33468144